CLINICAL TRIAL: NCT06611956
Title: Needs Assessment Among Carers of Someone With Suicidal Thoughts
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2024-0404
Record Dates: First submitted 2024-09-04; First posted 2024-09-25 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Suicide Prevention; Informal Caregivers
Keywords: needs assessment; informal caregivers; suicide
MeSH Terms: conditions — Suicide Prevention; Suicide | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention (observational study) — No intervention (observational study)

SUMMARY:
With this study the investigators would like to gain insight into the experienced needs carers of individuals with suicidal thoughts, who attempted suicide or who died by suicide. By carers the investigators mean everyone who knows/knew someone close to them who is thinking about suicide, attempted suicide or died by suicide. By mapping out these needs, the investigators hope to better support carers and develop/improve initiatives and tools.

The investigators examine this by means of an online one-time questionnaire. In this questionnaire the investigators ask the participants questions about what it is like to be a carer and what are some of the experienced needs, as well as experiences with existing initiatives/tools.

ELIGIBILITY:
Inclusion Criteria:

* 16 years or older
* Someone close to them has experienced suicidal thoughts, attempted suicide or died by suicide in the past three years
* Access to internet
* Understand sufficient Dutch (to complete the questionnaire)

Exclusion Criteria:

* /

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants are inidividuals (16 years or older) who know someone close to them with suicidal thoughts and/or behaviors in the past three years.
Sampling Method: Non-Probability Sample
Enrollment: 2255 (Actual)
Dates: Start 2024-11-29 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Background information: information on the participant | Baseline. Completing the questionnaire will take about 15-20 minutes
  Personal information (self-developed questionnaire): age, gender identity, education, cultural background, work status, recruitment type
Background information: information on the suicidal person | Baseline. Completing the questionnaire will take about 15-20 minutes
  Information on the suicidal person (self-developed questionnaire): relationship with the person, age, gender identity, suicidality, degree of contact
Experienced burden: suicidality | Baseline. Completing the questionnaire will take about 15-20 minutes
  based on national health survey (Sciensano, 2018)
Experienced burden when supporting the individual with suicdial thoughts | Baseline. Completing the questionnaire will take about 15-20 minutes
  self-developed questionnaire on the role of the carer and current degree of care
Experienced burden when supporting the individual with suicdial thoughts | Baseline. Completing the questionnaire will take about 15-20 minutes
  Zarit Caregiver Burden 4-item questionnaire (Zarit et al., 1985; Higginson et al., 2010)
Experienced burden: psychological stress | Baseline. Completing the questionnaire will take about 15-20 minutes
  Kessler Psychological Distress Scale , 6-item (Kessler et al., 2002, 2003)
Experienced needs | Baseline. Completing the questionnaire will take about 15-20 minutes
  Self-developed questionnaire examining the need for information, need for support and needs with regards to health care
Experience with existing initiatives and tools | Baseline. Completing the questionnaire will take about 15-20 minutes
  Self-developed questionnaire about the experience of participants with existing initiatives and tools

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, PhD, Principal Investigator — Flemish Centre of Expertise in Suicide Prevention (Ghent University)
Locations (1):
- Flemish Centre of Expertise in Suicide Prevention, Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No